CLINICAL TRIAL: NCT00292305
Title: Crush- or Culotte Stenting of Bifurcation Lesions Using Drug Eluting Stents? A Randomized Nordic Multicenter Study (BIF II)
Brief Title: Nordic Bifurcation Stent Technique Study (BIF II)
Acronym: BIF II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Cordis US Corp. (Industry)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, MD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050116
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: PCI; Bifurcation lesion
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention; Methods; Nerve Crush

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- T-crush stenting (Experimental): Percutaneous coronary intervention with implantation of a stent
  Interventions: Procedure: Percutaneous coronary intervention
- Culotte stenting (Active Comparator): Percutaneous coronary intervention with stent
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Implantation of coronary stent in bifurcation lesions
  Other Names: PCI; PTCA; Techniques; Crush; Culotte

SUMMARY:
This is a study of crush- or culotte stenting of bifurcation lesions using drug eluting stents. This is a randomized Nordic multicenter study including 400 patients with angina pectoris with clinical angiographic follow-up.

DETAILED DESCRIPTION:
Design:

* Randomized open multicentre trial.

Patients:

* Number 400.

Randomization:

* Treatment strategy culotte technique or T-crush stenting

Primary end-point:

* Combined end point of: cardiac death, myocardial infarction, stent thrombosis or TVR after 6 months.

Secondary end points

* Clinical
* MACE (cardiac death, MI, stent thrombosis or TVR) during hospital period, after 1 and 8 months.
* Cardiac death during hospital period, after 1, 6 and 8 months.
* Myocardial infarction during hospital period, after 1, 6 and 8 months.
* Stent thrombosis during hospital period, after 1, 6 and 8 months.
* TVR during hospital period, after 1, 6 and 8 months.
* Total death during hospital period, after 1, 6 and 8 months.
* TLR during hospital period, after 1, 6 and 8 months.
* Myocardial infarction related to index procedure.
* CCS-angina score after 6 and 8 months.
* Angiographic
* Late loss of main vessel and side branch after 8 months.
* Percentual diameter stenosis of main vessel and side branch after 8 months.
* Angiographic restenosis (> 50% diameter stenosis) rate of main vessel and side branch after 8 months.

End point evaluation:

* Primary and secondary end points will be assessed by an independent end point committee.
* The end point committee will consist of experienced interventional cardiologists.
* End point definitions:
* Q wave myocardial infarction. Appearance of a new Q wave in two or more contiguous leads on ECG.
* Non Q wave myocardial infarction. Infarction, which is considered present in a patient having clinical, angiographic, electrocardiographic, and/or laboratory evidence of myocardial necrosis with an ECG showing no new Q waves.

  * Procedure related myocardial infarction. A > threefold increase of CK-MB/or Troponin-T/I.
  * Target lesion revascularization. Coronary by-pass operation with grafting or PCI of index lesion.
  * Target vessel revascularization. Coronary by-pass operation with grafting or PCI of index vessel.
  * Stent thrombosis. Thrombotic occlusion of index stent/stents.
  * Vessel measurement. Proximal reference diameter: Vessel diameter proximal to lesion. Distal reference diameter: Vessel diameter distal to lesion. Reference diameter: Mean of proximal and distal vessel diameter. Percentual diameter stenosis: (Reference diameter - minimal luminal diameter)/reference diameter in percent.
  * Angiographic restenosis. > 50% diameter stenosis.

Angiographic core lab:

* The index and the follow-up angiograms will be assessed blindly by the QCA core lab at the Department of Cardiology, Skejby Hospital, 8200 Aarhus N, Denmark.

Definition of index angiography

* The angiography obtained during the PCI procedure will be used as index angiography.
* Follow-up angiography. After 8 months, conventional diagnostic angiography will be performed and the projections used at the index angiography will be repeated.

Steering committee

* The steering committee members will be selected on basis of participation in the study, see below. All steering committee members will have full access to the database and will participate in the interpretation of data.

Progress of the study

* The progress of the study will be checked on a weekly basis by the steering committee. They will receive and evaluate data on inclusion rate and the primary end point event rate. Further, the steering committee will receive and evaluate the weekly safety data on the rate of stent thrombosis in the three groups.

Statistics and Data Management

* The statistical analyses will be performed by UNI-C, University of Aarhus.
* Primary end point. The composite of the primary end points at six months follow-up will be analyzed by the Kaplan-Meier method. Differences between the event-free survival curves for the three groups will be compared with the use of the Wilcoxon and log-rank tests.
* Two-sided test is used, and the p-value considered to indicate significance will be 0.05.
* Secondary end points and other parameters: For continuous variables, differences between the treatment groups will be evaluated by analysis of variance or Wilcoxon's rank-sum test. For discrete variables, differences will be expressed as counts, and percentages will be analyzed with Fisher's exact test. Secondary end-points will be assessed after 8 months.
* Two-sided test is used, and the p-value considered to indicate significance will be 0.05.

Safety

* For safety reasons, stent thrombosis after one month will be monitored continuously. A stent thrombosis rate of > 5% in any of the treatment groups will necessitate premature termination of the trial.

Analysis Population

* Results are analyzed according to the intention-to-treat principle i.e. patients randomized to a certain group will be followed and assessed irrespectively of the actual treatment. Protocol violations will be noted and the responsible centers notified.

Sample size calculation

* 200 patients will be included in each group, with a total of 400 patients in the study. This is based on the following: We expect a MACE rate of 25% in the control group and 13% in the interventional group. With an alfa of 5% and a strength of 80%, 167 patients will be needed in each group (two-sided chi square test) to demonstrate this difference. By including 200 patients in each group, a possible dropout before follow-up is counted for.

Randomization procedure

* The patient will be randomized before insertion of any stent. Both main vessels and side branch may be wired and predilated before randomization.
* There will be a block randomization according to country, a stratification according to sex, age > 70 years, diabetes, use of GPIIb/IIIa blocker and +/- angiographic follow up.
* The patients will be computer randomized by a 24 hour telephone service. The PARAVOX system will be used.

Monitoring of the study

* Data will be monitored according to GCP rules by independent professionals. During the trial, the monitor will have regular contacts with the trial site(s), including visits to ensure that the trial is conducted and documented properly in compliance with the protocol, GCP and applicable regulatory requirements.

Publication

* Results will be published in an international cardiovascular journal. Publication and author issues will be decided by the steering committee on the basis of general involvement in the study (core lab. function, end point committee membership etc.) and on the number of included patients.

ELIGIBILITY:
Inclusion Criteria:

* Stable or unstable AP.
* Bifurcation lesion of "LAD/diagonal", "Cx/obtuse marginal", "RCA-PDA/posterolateral branch" or "LM/Cx/LAD".
* Diameter of main vessel by visual estimate > 3.0 mm.
* Diameter of side branch by visual estimate > 2.5 mm.
* Signed informed consent

Exclusion Criteria:

* ST-elevation AMI within 24 hours.
* Expected survival < 1 year.
* S-creatinine > 200 Umol/l.
* Allergy to aspirin, clopidogrel or ticlopidine.
* Allergy to sirolimus.
* Left main bifurcation in a non-right dominant system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2005-09; Primary Completion 2007-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Combined end point of: cardiac death, myocardial infarction, stent thrombosis or TVR | after 6 months

SECONDARY OUTCOMES:
Clinical MACE | December 2008
MACE (cardiac death, myocardial infarction, stent thrombosis or TVR) | during hospital period; after 1 and 8 months
Cardiac death | during hospital period; after 1, 6 and 8 months
Myocardial infarction | during hospital period; after 1, 6 and 8 months
Stent thrombosis | during hospital period; after 1, 6 and 8 months
TVR | during hospital period; after 1, 6 and 8 months
Total death | during hospital period; after 1, 6 and 8 months
TLR | during hospital period; after 1, 6 and 8 months
CCS-angina score | after 6 and 8 months
Late loss of main vessel and side branch | after 8 months
Percentual diameter stenosis of main vessel and side branch | after 8 months
Angiographic restenosis (> 50% diameter stenosis) rate of main vessel and side branch | after 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Leif Thuesen, MD, Study Director — Director Cardiac Cath. Lab, Skejby Hospital, University of Aarhus
Locations (1):
- Skejby Hospital, University of Aarhus, Aarhus, Denmark